CLINICAL TRIAL: NCT00773799
Title: Mastering Hospital Antimicrobial Resistance and Its Spread Into the Community
Acronym: MOSAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: yehuda carmeli, TASMC
Other Study IDs: TASMC-08-YC-239-CTIL
Record Dates: First submitted 2008-10-06; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: ESBL Infection; Methicillin-Resistant Staphylococcus Aureus
Keywords: To define activities and patient characteristics likely to lead to dissemination of resistant bacteria in rehabilitation centers and; To define specific risk factors for acquisition of resistant bacteria (ESBL producers and MRSA) in rehabilitation centers.; ESBL producers; MRSA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rehabilitation center's hospitalized patients

SUMMARY:
Data on occurrence of antimicrobial resistant bacteria acquisition in rehabilitation centers will be collected. After removal of patient identifiers, information regarding the patients population will be entered into electronic sheet. The phase will last twelve months in each center.

DETAILED DESCRIPTION:
All patients admitted to the department will be examined on admission, two weeks latter and monthly by obtaining nares and perirectal cultures. These cultures will be processed for detection the target organisms. This activity is part of the good medical practice and is performed on routine basis in various hospital units

Epidemiological data will be collected from patient records. This data will be stored after removal of all patients' identifiers. These data will be transferred for analysis to Tel Aviv Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients are older then 18 years old

Exclusion Criteria:

* Age 18 years or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A rehabilitation center's department in which the hospitalized patients are older then 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
A rehabilitation center's department in which the hospitalized patients are older then 18 years old. | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda carmeli, MD MPH, Principal Investigator — TASMC
Locations (1):
- Tasmc, Tel Aviv, Israel

REFERENCES:
- [Background] Vovko P, Retelj M, Cretnik TZ, Jutersek B, Harlander T, Kolman J, Gubina M. Risk factors for colonization with methicillin-resistant Staphylococcus aureus in a long-term-care facility in Slovenia. Infect Control Hosp Epidemiol. 2005 Feb;26(2):191-5. doi: 10.1086/502525. PMID 15756891
- [Background] Lucet JC, Grenet K, Armand-Lefevre L, Harnal M, Bouvet E, Regnier B, Andremont A. High prevalence of carriage of methicillin-resistant Staphylococcus aureus at hospital admission in elderly patients: implications for infection control strategies. Infect Control Hosp Epidemiol. 2005 Feb;26(2):121-6. doi: 10.1086/502514. PMID 15756880
- [Background] Ben-Ami R, Schwaber MJ, Navon-Venezia S, Schwartz D, Giladi M, Chmelnitsky I, Leavitt A, Carmeli Y. Influx of extended-spectrum beta-lactamase-producing enterobacteriaceae into the hospital. Clin Infect Dis. 2006 Apr 1;42(7):925-34. doi: 10.1086/500936. Epub 2006 Feb 27. PMID 16511754
- [Background] Stelfox HT, Bates DW, Redelmeier DA. Safety of patients isolated for infection control. JAMA. 2003 Oct 8;290(14):1899-905. doi: 10.1001/jama.290.14.1899. PMID 14532319
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Pope C, van Royen P, Baker R. Qualitative methods in research on healthcare quality. Qual Saf Health Care. 2002 Jun;11(2):148-52. doi: 10.1136/qhc.11.2.148. PMID 12448807
- [Background] Bartholomew LK, Parcel GS, Kok G. Intervention mapping: a process for developing theory- and evidence-based health education programs. Health Educ Behav. 1998 Oct;25(5):545-63. doi: 10.1177/109019819802500502. PMID 9768376
- [Background] van Bokhoven MA, Kok G, van der Weijden T. Designing a quality improvement intervention: a systematic approach. Qual Saf Health Care. 2003 Jun;12(3):215-20. doi: 10.1136/qhc.12.3.215. PMID 12792013
- [Background] Smith DL, Dushoff J, Perencevich EN, Harris AD, Levin SA. Persistent colonization and the spread of antibiotic resistance in nosocomial pathogens: resistance is a regional problem. Proc Natl Acad Sci U S A. 2004 Mar 9;101(10):3709-14. doi: 10.1073/pnas.0400456101. Epub 2004 Feb 25. PMID 14985511